CLINICAL TRIAL: NCT06070272
Title: Investigating the Dynamics of Patient Engagement and Trends in Participation in Recurrent Prostate Cancer Clinical Trials
Brief Title: Determining Patterns In Trial Experiences of Recurrent Prostate Cancer Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 72630763
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Prostate Cancer
Keywords: Recurrent Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical studies, with a dedicated focus on recurrent prostate cancer, play a pivotal role in evaluating the safety and effectiveness of novel treatments for this condition.

These trials serve as essential tools to determine whether new medications outperform traditional therapies, providing substantial evidence to endorse their broader utilization.

It will also try to analyze data from the perspective of different demographic groups to check for recurring trends which might yield insights for the sake of future patients with recurrent prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Diagnosis of recurrent prostate cancer
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Enrolled in another research study
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Inability to provide written informed consent

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients with recurrent prostate cancer who are actively considering enrolling in a clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to participate in a recurrent prostate cancer clinical research | 3 months
Rate of patients who remain in recurrent prostate cancer clinical research to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hefermehl LJ, Disteldorf D, Lehmann K. Acknowledging unreported problems with active surveillance for prostate cancer: a prospective single-centre observational study. BMJ Open. 2016 Feb 17;6(2):e010191. doi: 10.1136/bmjopen-2015-010191. PMID 26888730
- [Background] Wollersheim BM, Helweg E, Tillier CN, van Muilekom HAM, de Blok W, van der Poel HG, van Asselt KM, Boekhout AH. The role of routine follow-up visits of prostate cancer survivors in addressing supportive care and information needs: a qualitative observational study. Support Care Cancer. 2021 Nov;29(11):6449-6457. doi: 10.1007/s00520-021-06222-9. Epub 2021 Apr 26. PMID 33900459
- [Background] Ye D, Zhang W, Ma L, Du C, Xie L, Huang Y, Wei Q, Ye Z, Na Y. Adjuvant hormone therapy after radical prostatectomy in high-risk localized and locally advanced prostate cancer: First multicenter, observational study in China. Chin J Cancer Res. 2019 Jun;31(3):511-520. doi: 10.21147/j.issn.1000-9604.2019.03.13. PMID 31354220

DOCUMENTS (1):
  • Informed Consent Form (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT06070272/ICF_000.pdf